CLINICAL TRIAL: NCT03047252
Title: Home-based Rehabilitation With A Novel Digital Biofeedback System Versus Conventional Rehabilitation After Total Knee Replacement: a Feasibility Study
Brief Title: Rehabilitation for Total Knee Replacement: a Novel Biofeedback System Versus Conventional Home-based Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Collaborators: Hospital da Prelada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH-TKR-01
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Knee Osteoarthritis; Arthropathy of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All patients will be assessed for clinical outcomes by an independent rater blinded to the study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Home-based rehabilitation sessions performed with the novel digital biofeedback system.
  Patients will be instructed to perform exercise sessions in at least 5 days per week, but compliance to this schedule is not mandatory per protocol.
  Interventions: Device: Home-based rehabilitation with a digital biofeedback system
- Conventional rehabilitation group (Active Comparator): Home-based rehabilitation sessions provided by a Physical Therapist, 3 times a week for 8 weeks. Each session will have a duration of 60 minutes. Patients will be instructed to perform additional unsupervised sessions in at least two other days, but compliance to these extra sessions is not mandatory per protocol.
  Interventions: Other: Conventional Home-based rehabilitation

INTERVENTIONS:
Device: Home-based rehabilitation with a digital biofeedback system — The system will be used independently by the patients to perform rehabilitation sessions at home, under remote monitoring from the clinical team. A tailored rehabilitation program will be prescribed, based on the following principles:
  STAGE 1 (Weeks 0-2) Open kinetic chain exercises without added resistance: lying, sitting and standing (with support) Strengthening of hip flexors and extensors Ice pack application after each session and throughout the day as needed STAGE 2 (weeks 3-6) Open kinetic chain exercises with added resistance, progressing to closed kinetic chain exercises, with strengthening of knee flexors and extensors and knee stabilization Progression to standing exercises without support lying, sitting and standing (with support) Exercises with steps Ice pack application after each session and throughout the day as needed STAGE 3 (Weeks 7-8) Eccentric strengthening exercises Exercises involving steps Multi-directional exercises
  Other Names: SWORD Phoenix
  Arms: Experimental group
Other: Conventional Home-based rehabilitation — Patients will perform 3 weekly rehabilitation sessions, with a duration of 1 hour, for 8 weeks, provided by a physical therapist. The rehabilitation program will respect the following principles:
  STAGE 1 (Weeks 0-2) Soft tissue massage Active assisted mobilisation of the knee to increase range of motion Gait training with bilateral support Open kinetic chain exercises without added resistance Strengthening of hip flexors and extensors Ice pack application STAGE 2 (weeks 3-6) Soft tissue massage Active assisted mobilisation of the knee to increase range of motion Open kinetic chain exercises with added resistance, progressing to closed kinetic chain exercises, with strengthening of knee flexors/ extensors and knee stabilisation Gait training with progressive withdrawal of external support Ice pack application STAGE 3 (Weeks 7-8) Eccentric strengthening exercises Exercises involving steps Weight-bearing exercises on uneven surfaces Ice pack application
  Arms: Conventional rehabilitation group

SUMMARY:
The study was designed to test patient acceptance and system usability and to assess clinical outcomes of a home-based rehabilitation program using a novel kinematic biofeedback system in the rehabilitation after total knee replacement versus conventional rehabilitation, This system allows the patients to perform independent rehabilitation sessions at home, under remote monitoring from the clinical team.

The investigators hypothesize that the system will be well received by patients and that the clinical outcomes will be at least similar those of conventional rehabilitation.

This is a quasi-randomized controlled trial with active comparator. Patients will be enrolled pre-operatively and divided into 2 groups: experimental group and conventional rehabilitation group according to geographical criteria. Both groups will perform 8 weeks of rehabilitation starting between day 7 and 10 after surgery.

The experimental group will perform daily rehabilitation sessions at home using the system, under remote monitoring from a physical therapist. The conventional rehabilitation group will perform 1h rehabilitation sessions 3 times a week, at home, given by a physical therapist.

The following feasibility outcomes will be registered: enrollment rate, retention rate (drop-outs), compliance to the program, independence of use, need for therapist contact and patient satisfaction.

Clinical outcomes will be measured at weeks 4 and 8 and then at 3 and 6 months. The primary outcome will be measured in terms of patient performance in the Timed-up-and-Go (TUG) test in comparison with the pre-operative score. Secondary outcomes will be measured in terms of: b) Knee Osteoarthritis Outcome Score); c) range of motion of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Clinical and imaging evidence of knee osteoarthritis
* Indication for total knee replacement according to the patient´s orthopedic surgeon
* Ability to walk unaided, with unilateral or bilateral support
* Availability of a carer to assist the patient after surgery

Exclusion Criteria:

* Patients admitted for revision of total knee replacement
* Contralateral hip or knee osteoarthritis severely limiting patient mobility and ability to comply with a rehabilitation program
* Aphasia, dementia or psychiatric comorbidity interfering with the communication or compliance to the rehabilitation process
* Respiratory, cardiac, metabolic or other condition incompatible with at least 30 minutes of light to moderate physical activity
* Major medical complications occurring after surgery that prevent the discharge of the patient within 10 days after the surgery
* Other medical and/or surgical complications that prevent the patient from complying with a rehabilitation program
* Blind and/or illiterate patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-05-27 (Actual); Study Completion 2018-05-27 (Actual)

PRIMARY OUTCOMES:
Change in the Timed up And Go Test score | Baseline; 4 and 8 weeks after initiation of rehabilitation program and then at 3 and 6 months after surgery
  The timed up and go requires a patient to rise from a chair walk three meters around a piece of tape and return to the chair again as quickly as possible.

SECONDARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline; 4 and 8 weeks after initiation of rehabilitation program and then at 3 and 6 months after surgery
  The KOOS is a standardized and validated patient outcome score that assesses functional limitation in patient with knee problems.
Change in Knee Range of Motion (degrees) | Baseline; 4 and 8 weeks after initiation of rehabilitation program and then at 3 and 6 months after surgery
  Change in knee flexion/extension measured in degrees

OTHER OUTCOMES:
Enrollment rate | At the end of patient enrollment- up to 18 months after trial initiation
  This will be measured through the percentage of patients that actually enroll in the study after initial screening.
Retention rate | At week 8
  This will be assessed through the percentage of patients in the experimental group that complete the 8-week program
Independence of use | For each patient, at week 8 or upon dropout.
  This will be assessed through the percentage of patients in the experimental group that require the assistance of a caregiver in interacting with the system.
Compliance | For each patient, at week 8.
  This will be measured by calculating the percentage of patients allocated to the experimental group that performed at least 5 weekly sessions throughout the program
Patient Satisfaction | At week 8 or upon dropout.
  This will be measured in the experimental group by answering the following question: "On a scale from 0 to 10, how likely are you to recommend this intervention to a friend or neighbour?". Scores of 9 and 10 will be considered "good", 7 and 8 "neutral" and less than 7 "bad".

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — Sword Health, SA
Locations (1):
- Hospital da Prelada - Dr. Domingos Braga da Cruz, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made available in PDF format. Aggregate study results, with anonymised individual participant data will be made available in Excel format
Supporting Information: Study Protocol, SAP
Time Frame: Upon study publication, for at least five years.
Access Criteria: Study protocol is already available in clinicaltrials.gov and the excel file with the aggregate results will be made available upon study publication, for at least 5 years.

REFERENCES:
- [Derived] Correia FD, Nogueira A, Magalhaes I, Guimaraes J, Moreira M, Barradas I, Molinos M, Teixeira L, Tulha J, Seabra R, Lains J, Bento V. Medium-Term Outcomes of Digital Versus Conventional Home-Based Rehabilitation After Total Knee Arthroplasty: Prospective, Parallel-Group Feasibility Study. JMIR Rehabil Assist Technol. 2019 Feb 28;6(1):e13111. doi: 10.2196/13111. PMID 30816849